CLINICAL TRIAL: NCT03307980
Title: A FACTOR IX (FIX) GENE TRANSFER, MULTI CENTER EVALUATION OF THE LONG TERM SAFETY AND EFFICACY STUDY OF PF 06838435 AND A DOSE ESCALATION SUBSTUDY IN INDIVIDUALS WITH HEMOPHILIA B
Brief Title: Long-term Safety and Efficacy Study and Dose-Escalation Substudy of PF 06838435 in Individuals With Hemophilia B
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C0371003; SPK-9001-LTFU-101 (Other: Alias Study Number)
Record Dates: First submitted 2017-09-29; First posted 2017-10-12 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia B
Keywords: gene therapy; BeneGene LTE; hemophilia; SPK-9001; Factor IX; FIX
MeSH Terms: conditions — Hemophilia B; Hemophilia A

STUDY DESIGN:
Intervention Model Description: This study was originally designed as a long-term follow up study for individuals dosed in Study C0371005 to evaluate the overall long-term safety, durability of transgene expression, and effect on clinical outcomes of PF-06838435 mediated gene transfer. For these individuals this study will last for 5 years providing a minimum of 6 years of follow up post vector administration.
  Amendment 2 of this study introduces a dose-escalation substudy to evaluate the safety, tolerability, and kinetics of a single IV infusion of PF-06838435 at a higher dose(s) than that used in the C0371005 study. For these participants this study will last for a total of 6 years post vector administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-06838435 Dose-Escalation (Experimental): Single intravaneous infusion of PF-06838435. After 2 participants receive initial dose, data will be evaluated and a decision will be made to escalate or reduce the dose being evaluated, increase the number of participants receiving the dose, or stop dosing. Multiple iterations may be undertaken.
  Interventions: Biological: PF-06838435 (formerly SPK-9001)

INTERVENTIONS:
Biological: PF-06838435 (formerly SPK-9001) — Gene Therapy: A novel, bioengineered adeno-associated viral vector carrying human factor IX variant

SUMMARY:
Long-term safety and efficacy follow-up for participants with Hemophilia B who were previously treated in the C0371005 (formerly SPK-9001-101) study, and a dose-escalation sub-study evaluating safety, tolerability, and kinetics of a higher dose with long-term safety and efficacy follow-up. Participants in the substudy do not need to have participated in C0371005.

DETAILED DESCRIPTION:
Evaluation of the long-term level of persistence and potential late or delayed adverse events associated with PF-06838435 (formerly SPK-9001), assessment of the durability of the transgene expression, and determination of the effects of PF-06838435 on clinical outcomes in individuals who have previously received a single administration of PF-06838435 in the C0371005 study. Amendment 2 of this study incorporates a dose-escalation substudy to evaluate the safety, tolerability, and kinetics of a single IV infusion of PF-06838435 at a higher dose than that used in the C0371005 study. The dose-escalation participants will also be followed for long-term safety and efficacy.

ELIGIBILITY:
This study is currently only enrolling into the dose-escalation substudy with subsequent long-term follow-up. The Eligibility Criteria for entry into the dose-escalation substudy is presented below:

Inclusion Criteria:

1. Able to provide informed consent and comply with requirements of the study
2. Males age 18 to 65 years with confirmed diagnosis of hemophilia B (≤2 IU/dL or ≤2% endogenous factor IX)
3. Received ≥50 exposure days to factor IX products
4. No measurable factor IX inhibitor as assessed by the central laboratory and have no prior history of inhibitors to factor IX protein
5. Agree to refrain from donating sperm and either abstain from intercourse or use reliable barrier contraception until 3 consecutive semen samples are negative for vector sequences

Exclusion Criteria:

1. Evidence of active hepatitis B or C
2. Currently on antiviral therapy for hepatitis B or C
3. Have significant underlying liver disease
4. Serological evidence* of HIV-1 or HIV-2 with CD4 counts ≤200/mm3 (* participants who are HIV+ and stable with CD4 count >200/mm3 and undetectable viral load are eligible to enroll)
5. Neutralizing antibody titers to the capsid portion of PF-06838435 above the established threshold
6. Sensitivity to heparin or heparin induced thrombocytopenia; sensitivity to any of the study interventions, or components thereof, or drug or other allergy
7. Previously dosed in a gene therapy research trial at any time or in an interventional clinical study within 3 months of screening visit
8. Any concurrent clinically significant major disease or condition
9. Unable or unwilling to comply with the study procedures

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Genetic males
Enrollment: 21 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2029-06-08 (Estimated); Study Completion 2029-06-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of PF-06838435 related adverse events | Baseline up to Year 6

SECONDARY OUTCOMES:
Incidence of clinically significant changes from baseline | Baseline up to 52 weeks
  Clinically significant changes in physical examination, vital signs, laboratory values. (to be reported as AEs, regardless of causality)
Incidence of protocol-defined medically important events | Baseline up to 52 weeks
  Clinical thrombotic events, FIX inhibitor development as assessed by Nijmegen Bethesda assay, Hypersensitivity reaction (eg, bronchospasm and anaphylaxis), Hepatic malignancy, Study intervention-related elevated hepatic transaminases that fail to improve or resolve, Malignancy assessed as having reasonable possibility of being related to study intervention (to be reported as SAEs).
Immune response against AAV capsid protein and hFIX transgene | Baseline up to 52 weeks
  Positive immune response based on peripheral blood mononuclear cell (PBMC) results by interferon gamma enzyme-linked immunospot assay (ELISPOT).
Coagulation Clotting Assay for FIX activity levels | Baseline up to Year 6
  Coagulation Clotting assays to assess FIX activity levels (percent of normal)
Mean and standard deviation of vector-derived FIX Activity levels | Baseline up to 52 weeks
  Mean and standard deviation of peak and steady-state FIX Activity
Mean and standard deviation of FIX Antigen levels | Baseline up to 52 weeks
  Mean and standard deviation of FIX Antigen levels
Annualized bleeding rate (ABR) | Baseline up to Year 6
  ABR (not including those for surgery)
Annualized (factor FIX) infusion rate | Baseline up to Year 6
  AIR (not including those for surgery)
Total factor consumption (IU) | Baseline up to Year 6
  total quantity of factor infused annually (not including those for surgery) as recorded on the infusion log
Total number of bleeding events | Baseline up to Year 6
  spontaneous and traumatic
Haem-A-QoL | Baseline up to Year 6
  Quality-of-life (QoL) assessment
EQ-5D-5L | Baseline up to Year 6
  Quality-of-life (QoL) assessment
Brief Pain Inventory | Year 2 up to Year 6
  Quality-of-life (QoL) assessment
McGill Pain Questionnaire | Baseline up to 52 weeks
  Quality-of-life (QoL) assessment

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (17):
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - UC Davis Ellison Ambulatory Care Clinic, Sacramento, California
  - UC Davis Medical Center department of Radiology, Sacramento, California
  - UC Davis Medical Center, Sacramento, California
  - UC Davis Midtown Cancer Center, Sacramento, California
  - UC DavisHealth Main Hospital, Sacramento, California
  - LA Center for Bleeding and Clotting Disorders - Metairie, Metairie, Louisiana
  - Tulane Lakeside Hospital, Metairie, Louisiana
  - LA Center for Bleeding and Clotting Disorders, New Orleans, Louisiana
  - Tulane University Clinical Translational Unit, New Orleans, Louisiana
  - Tulane University Hospitals and Clinic, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Louisiana Center for Advanced Medicine, Slidell, Louisiana
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Weill Cornell Medicine - New York Presbyterian Hospital, New York, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia
- Canada (2):
  - McMaster University Medical Centre - Hamilton Health Sciences, Hamilton, Ontario
  - McGill University Health Center - Research Institute, Montreal, Quebec
- Turkey (Türkiye) (2):
  - Istanbul Universitesi Onkoloji Enstitusu Çocuk Hematoloji Onkoloji Bilim Dali, Istanbul
  - Ege Universitesi Tip Fakultesi Cocuk Sagligi ve Hastaliklari Anabilim Dali, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Wojciechowski J, Gaitonde P, Hughes JH, Ravva P. Population Modeling of Factor IX Activity Following Administration of Fidanacogene Elaparvovec Gene Therapy in Participants with Hemophilia B. Clin Pharmacokinet. 2025 Oct;64(10):1531-1548. doi: 10.1007/s40262-025-01535-y. Epub 2025 Aug 1. PMID 40750723
- [Derived] Rasko JEJ, Samelson-Jones BJ, George LA, Giermasz A, Ducore JM, Teitel JM, McGuinn CE, High KA, de Jong YP, Chhabra A, O'Brien A, Smith LM, Winburn I, Rupon J. Fidanacogene Elaparvovec for Hemophilia B - A Multiyear Follow-up Study. N Engl J Med. 2025 Apr 17;392(15):1508-1517. doi: 10.1056/NEJMoa2307159. PMID 40239068
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0371003